CLINICAL TRIAL: NCT00436436
Title: A Phase 2 Study of O-Benzylguanine (O-BG) and Temozolomide in Patients With Glioblastoma Progressing at Least 3 Months After Completion of Primary Treatment With Radiation Therapy and Temozolomide
Brief Title: O(6)-Benzylguanine and Temozolomide in Treating Patients With Glioblastoma Multiforme That Did Not Respond to Previous Temozolomide and Radiation Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed to accrual after the company chose to stop development of the drug.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark Gilbert, M.D., Branch Chief, Neuro-Oncology Branch, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070052; NCI-07-C-0052; AOI-NCI-07-C-0052; CDR0000529875 (Other: nci)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult gliosarcoma; recurrent adult brain tumor; adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — O(6)-benzylguanine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- O6-benzylguanine & Temozolomide in Glioblastoma (Experimental): Patients receive O6-benzylguanine intravenous over 1 hour and oral temozolomide once daily on days 1-5. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: O6-benzylguanine; Drug: temozolomide

INTERVENTIONS:
Drug: O6-benzylguanine
  Other Names: 06-BG
Drug: temozolomide
  Other Names: Temodar

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as O(6)-benzylguanine and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving O(6)-benzylguanine together with temozolomide works in treating patients with glioblastoma multiforme that did not respond to previous temozolomide and radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of O6-benzylguanine and temozolomide in patients with temozolomide-resistant methylguanine methyltransferase-positive or -negative glioblastoma multiforme previously treated with radiotherapy.
* Determine, preliminarily, the toxicity of this regimen in these patients.

OUTLINE: Patients receive O6-benzylguanine intravenous (IV) over 1 hour and oral temozolomide once daily on days 1-5. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for at least 6 months.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme (GBM), including the following:

  * Small or large cell GBM
  * Gliosarcoma
* Temozolomide-resistant disease, as defined by the following:

  * Unequivocal evidence of tumor progression after receiving adjuvant temozolomide therapy for 5 consecutive days every 28 days for ≥ 2 courses
* Must have failed prior radiotherapy

  * Progression must be documented by MRI (while on a stable steroid dose for ≥ 5 days) ≥ 12 weeks after completion of radiotherapy
* Must have paraffin-embedded tissue blocks or ≥ 4 unstained paraffin-embedded microscope slides available from diagnosis

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Life expectancy > 8 weeks
* White blood cell (WBC) ≥ 3,000/mm(³)
* Absolute neutrophil count ≥ 1,500/mm(³)
* Platelet count ≥ 100,000/mm(³)
* Hemoglobin ≥ 10 g/dL (transfusion allowed)
* Aspartate aminotransaminase (AST) < 2 times upper limit of normal (ULN)
* Bilirubin < 2 times ULN
* Creatinine < 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* No significant medical illness that, in the opinion of the investigator, would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant active cardiac, hepatic, renal, or psychiatric disease
* No other known active malignancy except for nonmelanoma skin cancer or carcinoma in situ of the cervix
* No active infection requiring intravenous (IV) antibiotics
* No disease that would obscure toxicity or alter drug metabolism

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior temozolomide
* Prior resection of recurrent or progressive tumor allowed if all the following criteria are met:

  * Recovered from prior surgery
  * Residual disease after resection of recurrent tumor by computed tomography (CT) scan or magnetic resonance imaging (MRI) (while on a stable steroid dose for ≥ 5 days) ≤ 96 hours OR ≥ 4 weeks after surgery
* At least 12 weeks since prior radiotherapy
* No other prior therapy (i.e., polifeprosan 20 with carmustine implant [Gliadel wafers] or nitrosoureas)
* No other concurrent chemotherapy, radiotherapy, immunotherapy, or investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-11-13 (Actual); Primary Completion 2010-03-15 (Actual); Study Completion 2010-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard A Fine, M.D., Principal Investigator — NCI - Neuro-Oncology Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - NCI - Neuro-Oncology Branch, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- O6-benzylguanine & Temozolomide in Glioblastoma: Patients receive O6-benzylguanine intravenous over 1 hour and oral temozolomide once daily on days 1-5. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  O6-benzylguanine
  temozolomide
Period: Overall Study
Arm/Group | O6-benzylguanine & Temozolomide in Glioblastoma
Started | 12
Completed | 0
Not Completed | 12
Not completed — Progression | 4
Not completed — Adverse Event | 2
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | O6-benzylguanine & Temozolomide in Glioblastoma
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.03 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Best Objective Tumor Response Rate (Complete or Partial Response) in Patients With Methylguanine Methyltransferase (MGMT)-Positive Tumors as Assessed by Immunohistochemistry (IHC)
Description: The date of response will be the date the response is first radiographically documented following initiation of therapy (typically, the date of the actual imaging modality). Complete response is complete disappearance of all measurable and evaluable disease. No new lesions. No evidence of non-evaluable disease. Partial response is greater than or equal to a 50% decrease compared to baseline in the sum of products of perpendicular diameters of all measurable lesions.
Time Frame: 2-4 weeks
Population: No analysis was performed. The study was closed to accrual after the company chose to stop the development of the drug.
Arm/Group | O6-benzylguanine & Temozolomide in Glioblastoma
Number analyzed (Participants) | 0

2. Secondary Outcome: Objective Tumor Response Rate in Patients With Methylguanine Methyltransferase (MGMT)-Negative Tumors as Assessed by Immunohistochemistry (IHC)
Description: The date of response will be the date the response is first radiographically documented following initiation of therapy (typically, the date of the actual imaging modality). Complete response is complete disappearance of all measurable and evaluable disease. No new lesions. No evidence of non-evaluable disease. Partial response is greater than or equal to a 50% decrease compared to baseline in the sum of products of perpendicular diameters of all measurable lesions. Stable/No disease does not qualify for CR, PR, or progression. Progression is a 25% increase in the sum of products of all measurable lesions (or two largest lesions if too numerous) over the smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: 2-4 weeks
Population: Twelve patients were enrolled. The principal investigator wished to analyze the data but felt that there was insufficient data to report on and therefore closed the protocol when he left the National Cancer Institute (NCI).
Arm/Group | O6-benzylguanine & Temozolomide in Glioblastoma
Number analyzed (Participants) | 0

3. Secondary Outcome: Toxicity as Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v 3)
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module. Adverse events were assessed by the Common Terminology Criteria in Adverse Events (CTCAE)v3.
Time Frame: 18 months and 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | O6-benzylguanine & Temozolomide in Glioblastoma
Number analyzed (Participants) | 12
Participants | 12

4. Secondary Outcome: Best Overall Response
Description: Defined as the best tumor response recorded from the start of treatment until disease progression or withdrawal from the study. Complete response is complete disappearance of all measurable and evaluable disease. No new lesions. No evidence of non-evaluable disease. Partial response is greater than or equal to a 50% decrease compared to baseline in the sum of products of perpendicular diameters of all measurable lesions. Stable/No disease does not qualify for CR, PR, or progression. Progression is a 25% increase in the sum of products of all measurable lesions (or two largest lesions if too numerous) over the smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer
Time Frame: up to 2 years
Population: No analysis was performed. The study was closed to accrual after the company chose to stop the development of the drug.
Arm/Group | O6-benzylguanine & Temozolomide in Glioblastoma
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-free Survival
Description: Defined as the interval between the day of first administration of treatment and the first documentation of progressive disease or date of death. Progression is a 25% increase in the sum of products of all measurable lesions (or two largest lesions if too numerous) over the smallest sum observed (over baseline if no decrease) using the same techniques as baseline, OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer
Time Frame: up to 2 years
Population: No analysis was performed. The study was closed to accrual after the company chose to stop the development of the drug.
Arm/Group | O6-benzylguanine & Temozolomide in Glioblastoma
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival
Description: Defined as the interval between the day of first administration of treatment and the date of death.
Time Frame: up to 2 years
Population: No analysis was performed. The study was closed to accrual after the company chose to stop the development of the drug.
Arm/Group | O6-benzylguanine & Temozolomide in Glioblastoma
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 18 months and 4 days
Arm/Group | O6-benzylguanine & Temozolomide in Glioblastoma
All-Cause Mortality (participants affected / at risk) | 6/12
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | O6-benzylguanine & Temozolomide in Glioblastoma (N=12)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 2 (3)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (6)
Lymphopenia (Blood and lymphatic system disorders) | 2 (5)
Muscle weakness, generalized or specific area (not due to neuropathy)::Left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (3)
Platelets (Blood and lymphatic system disorders) | 3 (7)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Seizure (Nervous system disorders) | 4 (6)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
Death due to progressive disease (General disorders) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | O6-benzylguanine & Temozolomide in Glioblastoma (N=12)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 3 (4)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 2 (2)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (1)
Blood/Bone Marrow - Other (Specify, leukopenia) (Blood and lymphatic system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 2 (2)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 5 (7)
Lymphopenia (Blood and lymphatic system disorders) | 4 (5)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5 (8)
Platelets (Blood and lymphatic system disorders) | 4 (8)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Dr. Howard A. Fine is no longer with the National Cancer Institute (NCI). For historical reasons, he is listed as the (original principal investigator) study official for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No